CLINICAL TRIAL: NCT03446469
Title: Influence of Fascial Manipulation on Postural Sway and Ankle Range of Motion in Participants With Chronic Ankle Instability
Brief Title: Influence of Fascial Manipulation on Postural Sway and Ankle Range of Motion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manipal University (Other)
Responsible Party: Principal Investigator, Neha C. Kamani, Postgraduate student, Manipal University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ManipalU; CTRI/2018/02/011762 (Registry Identifier: Clinical Trials Registry - India)
Record Dates: First submitted 2018-01-23; First posted 2018-02-26 (Actual); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Ankle Injuries and Disorders : Chronic Ankle Instability
Keywords: Chronic ankle instability; Functional instability; Ankle sprain; postural sway; Fascial Manipulation
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Individuals with Chronic Ankle instability (Experimental): Individuals with history of ankle sprains will be screened using the inclusion criteria before being included in the study
  Interventions: Other: Fascial Manipulation

INTERVENTIONS:
Other: Fascial Manipulation — Myofascial release of densified centers of coordination

SUMMARY:
Fascia is defined as the soft tissue component of the connective tissue system. It is a continuous mesh that has several functions such as maintaining structural integrity and providing support and protection. Ligaments are part of the dense connective tissue system.

Studies conducted for ankle retinacula, which are thickened bands of fascia, also confirmed the presence of nervous tissue and proprioceptors within. Specific changes are seen in the MRI of ankle retinacula of individuals with chronic ankle instability. These changes include thickening of subcutaneous tissue. These structural changes may be responsible for interrupting the signals from the mechanoreceptors or also in damaging them.

Since fascial manipulation can help reduce the densifications of deep fascia, it is possible that on restoring the original structural and material properties, the proprioception may improve due to clearer signals from the mechanoreceptors. For a normal individual, recurrent sprains may lead to occupational absence and difficulty with their ADLs. Hence, there is a need for this study to determine the influence of FM on chronic ankle instability.

DETAILED DESCRIPTION:
Chronic ankle instability (CAI) is defined as "repetitive bouts of lateral ankle instability due to the sprain of the lateral collateral ligament of the ankle, resulting in numerous ankle sprains, episodes of giving way and decreased physical activity.

Individuals with chronic ankle instability often complain of repeated turning of the ankle especially on uneven surfaces, self-reported feelings of the ankle feeling wobbly way and a past history of at least one severe lateral ankle sprain.

The recurrence of ankle sprains can be attributed to the proprioceptive deficits that occur due to joint deafferentation. Freeman et al originally proposed that joint deafferentation is the loss of sensory input from the articular mechanoreceptors located in the capsule and ligaments of the affected joint. Proprioceptive deficits manifest in the form of impaired balance and postural control.

The objective of the study is to determine the effectiveness of fascial manipulation on improving ankle instability by measuring pre- and post-intervention measures of postural sway and ankle range of motion.

Luigi Stecco's biomechanical model acts as the foundation for describing the framework of the fascial system. This model describes a myofascial unit (MFU) as the functional unit of this system. A myofascial unit consists of unidirectional muscle fibers, fascia, nerve structures and other retinacular structures such as joint capsules and ligaments. Two crucial points can be identified along a myofascial unit. These points are known as the centre of perception (CP) and centre of coordination (CC). A total of six myofascial units have been established for each body segment and it is in these myofascial units that dysfunction will be seen. The indication or exhibition of these dysfunctions varies from one individual to the next. However, the etiology remains universal i.e. densification of the CC due to abnormal tensile and mechanical stresses. Movement and palpation assessments are carried out to identify the involved CCs which are focused on during treatment using fascial manipulation.

ELIGIBILITY:
Inclusion Criteria:

* Cumberland ankle instability score ≤27
* Subjective feeling of giving way of the ankle
* No history of acute injuries
* Previous history of ankle sprain

Exclusion Criteria:

* Lower limb surgery
* Neurological disorders with balance impairments (e.g. Parkinson's disease, Alzheimer's disease, stroke, multiple sclerosis)
* Known history of Diagnosed diabetic neuropathy
* Vestibular balance disorders
* Deformities of the foot
* History of acute ankle sprain
* Skin lesions localized to the affected lower limb

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2018-04-15 (Actual); Study Completion 2018-04-19 (Actual)

PRIMARY OUTCOMES:
Center of pressure (COP) velocity | 30 seconds
  COP velocity represents total distance traveled by the COP over time.
Center of pressure excursion | 30 seconds
  COP excursion represents the total distance traveled by the COP over the course of the trial duration

SECONDARY OUTCOMES:
Ankle dorsiflexion range of motion | 1 week
  Amount of flexion that can occur at the ankle joint in a weight bearing lunge starting from a neutral position
Foot and Ankle Disability Index (FADI) questionnaire | 1 week
  Subjective questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Sports Science, Medicine and Research, Udupi, Karnataka, India

IPD SHARING:
Plan to Share IPD: Undecided